CLINICAL TRIAL: NCT06589843
Title: Artificial Intelligent Image Processing and Diagnosis of Pulmonary Vessels in CT
Status: Not yet recruiting | Type: Observational
Sponsor: Xin Lou (Other)
Responsible Party: Sponsor-Investigator, Xin Lou, Chairman, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: NCCT-CTPA AI
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Radiology; Vascular Diseases
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Deep learning imaging enhancement — Conventional imaging or down-sampling imaging from CT or MR are enhanced by approved deep learning method.

SUMMARY:
In this study, patients with chest pain, lung cancer, pulmonary embolism, and routine inpatient physical examination were selected as the research objects, and the experimental design of retrospective cohort study was adopted to carry out artificial intelligence analysis related to pulmonary vascular diseases in patients with multi-dimensional big data. The multi-modal CT acquisition process included plain scan CT(NCCT) and CT pulmonary angiography (CTPA). Ctpa-like image effects can be simulated or reconstructed by non-enhanced plain scan CT images, so that CTPA-like image quality can be obtained without injecting contrast agent. The synthetic CTPA images were further analyzed by artificial intelligence to assist doctors in the intelligent diagnosis of pulmonary vascular diseases.

DETAILED DESCRIPTION:
A non-enhanced plain scan CT image simulates or reconstructs an image effect similar to that of CTPA through the following technical solutions:

1. Data acquisition: Obtain plain scan CT image data of the examined person, including multiple layers of image slices.
2. Image preprocessing: Preprocessing of plain scan CT images, including denoising, enhancing contrast and other steps, to improve image quality and lay the foundation for subsequent processing.
3. Vascular segmentation: Advanced image segmentation algorithms, such as the deep learning-based segmentation method, are used to segment the vascular structure from the preprocessed plain scan CT images. The key to this step is to accurately identify and extract vascular areas while reducing interference from non-vascular tissue.
4. Blood vessel enhancement: For the segmented blood vessel structure, a specific image enhancement algorithm is used to enhance blood vessels to make them clearer and more continuous.
5. Image synthesis: The enhanced vascular image is fused with the original plain scan CT image to generate the final CTPA image. During the synthesis process, the contrast between blood vessels and surrounding tissues can be adjusted as needed to optimize the display effect.
6. Post-processing and evaluation: Post-processing of synthesized CTPA images, such as smoothing, artifact removal, etc., and quality assessment to ensure that the images meet the needs of clinical diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18≤100 years old Scan the pulmonary artery and its major branches Patients with suspected pulmonary embolism who received CTPA had a set of CTPA and CT scans The image quality meets the requirements of diagnosis and post-processing Patients who completed the examination in accordance with the data collection criteria Clinical data and follow-up were complete

Exclusion Criteria:

* Age <18 years or age >100 years The image is incomplete or incorrect Pulmonary artery absent or underenhanced Severe motion artifacts or image noise affect evaluation of pulmonary embolism History of aortic reconstruction, replacement, or stent implantation Congenital variations in the whole or important branches of the aorta in adults (e.g. bovine aortic arch, abnormal right subclavian artery) Severe hypovolemia and hemodynamic instability Severe heart failure with low ejection fraction Dialysis patient

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chest pain, lung cancer, pulmonary embolism, and routine inpatient physical examination were studied
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2024-09-10 (Estimated); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
The performance of deep enhanced imaging in lesion detection and diagnosis | 2 year
  The performance of deep enhanced imaging in lesion detection and diagnosis, including imaging quality, accuracy, sensitivity and specificity in lesion detection and imaging diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Lou, Study Chair — Chinese PLA General Hospital